CLINICAL TRIAL: NCT05219136
Title: Improve the Comfort, Safety and Quality of Upper Endoscopy by a Modified Fasting Protocol：a Double-center, Prospective, Controlled Study
Brief Title: Improve the Comfort, Safety and Quality of Upper Endoscopy by a Modified Fasting Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The Affiliated Traditional Chinese Medicine Hospital Of Southwest Medical University (Unknown)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Fasting time
Record Dates: First submitted 2021-12-20; First posted 2022-02-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Gastroscopy; Feelings; Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Fasting Group (Active Comparator): In this parallel group, subjects are performed a conventional fasting protocol which requires 6-8h fasting for solid, 2h for clear liquids.
  Interventions: Other: Conventional Fasting Group
- Modified Fasting Group (Experimental): In this test group, a new protocol of 4h fasting for rice porridge, 2h for clear liquids is applied to subjects.
  The rice porridge is commercially available (New Rice Porridge®, Charm Kitchen Food Co., Ltd., Q/NBBD0001S). The volume is 300ml, with the energy as 105kJ per 100g, and it can be eaten after being heated or at room temperature.
  Interventions: Other: Modified Fasting Group

INTERVENTIONS:
Other: Modified Fasting Group — a new fasting protocol is applied to subjects.
  Arms: Modified Fasting Group
Other: Conventional Fasting Group — a conventional fasting protocol is applied to subjects.
  Arms: Conventional Fasting Group

SUMMARY:
This double-center, prospective, interventional study aims to include 200 gastroscopic procedures and investigate the relationship between fasting time and feeling of subjects. The subjects will all receive examination between 10:30 to 11:30am. In the control group, the subjects are required to start the fast at 10:00pm the day before examination and can not drink water after 8:00am on the day of examination. In the test group, the subjects are required to have customized rice congee before 6:30am on the examination day and can not drink water after 8:00am. All subjects complete questionnaire which include discomfort and willingness to accept the same fasting regimen.

ELIGIBILITY:
Inclusion Criteria:

* No history of benign and malignant tumors (including carcinoma and adenoma) of upper GI (including esophagus, stomach and duodenum)

Exclusion Criteria:

* Subjects that cannot stand the gastroscopy procedure or cannot cooperate with endoscopists
* Emergency endoscopy and therapeutic endoscopy
* Subjects with history of esophageal or stomach surgery or endoscopic surgery
* Pregnant
* Subjects that refuse to cooperate with data collection or sign the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
subject's discomfort | up to 1 week
  The feeling of the subject during the examination. 1) the score of mucosal restriction observed under gastroscope 2）the score of discomfort before gastroscopy 3）the score of discomfort during gastroscopy process. The discomfort feeling indicator was obtained from subject through a VAS scale. The score of mucosal restriction was obtained from endoscopists.

SECONDARY OUTCOMES:
incidence of adverse events | up to 1 week
  number of gastroscopy procedures with adverse event divided by the number of all gastroscopy procedures

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xin, Dr, Principal Investigator — Changhai Hospital; Luo-wei Wang, PhD, Study Chair — Changhai Hospital; Li Li, Dr, Principal Investigator — The Affiliated Traditional Chinese Medicine Hospital Of Southwest Medical University
Locations (2):
- China (2):
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - The Affiliated Traditional Chinese Medicine Hospital Of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No